CLINICAL TRIAL: NCT01838954
Title: The Effect of Short-wave Diathermy in Patients With Osteoarthritis of the Hand: A Randomized, Double Blinded, Placebo Controlled Trial
Brief Title: Short-wave Diathermy in Patients With Osteoarthritis of the Hand
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Medical University of Vienna (Other)
Responsible Party: Principal Investigator, Klaus Bobacz, principal investigator, Medical University of Vienna
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: MUW-1281571
Record Dates: First submitted 2013-04-16; First posted 2013-04-24 (Estimated); Last update posted 2015-04-10 (Estimated); Status verified 2015-04

CONDITIONS: Hand Osteoarthritis
Keywords: hand osteoarthritis; short-wave diathermy

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Short-wave diathermy (Active Comparator): Short-wave diathermy device turned on
  Interventions: Device: Short-wave diathermy
- control (Placebo Comparator): Short-wave diathermy device turned off

INTERVENTIONS:
Device: Short-wave diathermy — Device operating at a frequency of 27.12 MHz in continuous mode with an effective nominal output of 400 W in the patient circuit.
  Other Names: Ultratherm (Siemens) model 808i
  Arms: Short-wave diathermy

SUMMARY:
Due to constant strain the joints of the hands are frequently affected by osteoarthritis (OA).

Short-wave diathermy (SWD) is a form of electromagnetic therapy, which causes movement of ions, distortion of molecules, and creation of eddy currents and as a result heat is produced in deep tissue. Its claimed mechanism of action includes inducing an anti-inflammatory response, reducing joint stiffness, stimulating connective tissue repair, and reducing muscle spasm and pain.

Since the available studies were performed to study the large weight-bearing joints only, there is a lack in scientific evidence for the efficacy of SWD in hand OA.

The aim of this randomized, double blind, placebo-controlled study is to evaluate the effect of SWD on:

joint function in patients with hand OA. joint pain in patients with hand OA. grip strength in patients with hand OA. quality of live in patients with hand OA.

ELIGIBILITY:
Inclusion Criteria:

* Males and females > 18 years of age. All subjects who are not surgically sterile or postmenopausal must agree and commit to the use of a reliable method of birth control for the duration of the study.
* Persistent or transient pain/aching/stiffness in at least one DIP and/or PIP joint with or without bony swelling
* Hand X-ray showing alterations typical for OA
* If NSAIDs are used to treat finger joint pain dosage must be stable for at least 4 weeks
* Able and willing to give written informed consent and to comply with the requirements of the study protocol.

Exclusion Criteria:

* Prior treatment with any investigational agent within 30 days, or five half lives of the product, whichever is longer.
* Patients suffering from chronic inflammatory rheumatic disease (e.g. rheumatoid arthritis or positive rheumatoid factor or positive anti-CCP antibodies, seronegative spondylarthropathy, haemochromatosis, gout, chondrocalcinosis or other auto-immune diseases
* Stable dosage for at least 3 months with chondroitin sulfate, glucosamine, biphosphonate, corticosteroids, tetracyclines and estrogens is allowed.
* Prior use of any immunomodulating drug with possible effects on pro-inflammatory cytokine metabolism within 90 days a.o. corticosteroids, methotrexate, sulfasalazine, leflunomide, d-penicillamin, anti-malarials, cytotoxic drugs, TNF blocking agents
* If the patient is of child-bearing age, he/she must use effective means of contraception during the study.
* Use of anticoagulants (cumarins or low-molecular-weight-heparins)
* Subjects with hand OA showing or having suffered from transient inflammatory attacks of the IPJs characteristic for what has been termed 'inflammatory' or 'erosive' hand OA.
* Patient who has a known blood coagulation disorder
* metall implants (such as joint endoprothesis, pace-maker, implantable cardioverter/defibrillator, stents), piercings have to be removed prior to SWD treatment
* History of cancer or lymphoproliferative disease
* Comorbidities: uncontrolled diabetes, unstable ischemic heart disease, congestive heart failure (NYHA III, IV), recent stroke (within three months), uncontrolled hypertension (defined as screening systolic blood pressure > 160 mmHg or screening diastolic blood pressure > 100 mmHg), severe pulmonary disease requiring hospitalization or supplemental oxygen
* Persistent or recurrent infections or severe infections requiring hospitalization or treatment with iv antibiotics within 30 days, or oral antibiotics within 14 days prior to enrollment.
* Female subjects who are breast-feeding.
* History of clinically significant drug or alcohol abuse in the last year.
* Medical history of systemic lupus erythematosus or other connective tissue disease, RA, reactive arthritis, psoriasis
* Latex sensitivity.
* Reasonable expectation that the subject will not be able to satisfactorily complete the study. History of or current psychiatric illness, alcohol or drug abuse that would interfere with the subject's ability to comply with protocol requirements or give informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2012-03; Primary Completion 2016-04 (Estimated); Study Completion 2016-09 (Estimated)

PRIMARY OUTCOMES:
change in joint function in patients with hand OA (baseline, week 4 follow-up and week 12 follow-up) | week 0, week 4, week 12

SECONDARY OUTCOMES:
change in joint pain in patients with hand OA (baseline, week 4 follow-up and week 12 follow-up) | week 0, week 4, week 12
change in grip strength in patients with hand OA (baseline, week 4 follow-up and week 12 follow-up) | week 0, week 4, week 12
quality of live in patients with hand OA (baseline, week 4 follow-up and week 12 follow-up) | week 0, week 4, week 12

CONTACTS AND LOCATIONS:
Overall Officials: Klaus Bobacz, MD, Principal Investigator — Medical University of Vienna
Locations (1):
- Department of Internal Medicine III, Division of Rheumatology, Medical University of Vienna, Vienna, Vienna, Austria